CLINICAL TRIAL: NCT02540278
Title: Evaluation of the Positive Prevention PLUS Program Teen Pregnancy Prevention Program
Brief Title: Evaluation of the Positive Prevention PLUS Program
Acronym: PP+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California State University, San Bernardino (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Principal Investigator, Robert G. LaChausse, Principal Investigator, California State University, San Bernardino
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 09-149-1-5
Record Dates: First submitted 2015-08-25; First posted 2015-09-03 (Estimated); Last update posted 2015-09-03 (Estimated); Status verified 2015-09

CONDITIONS: Pregnancy in Adolescence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): Received the 11 lesson Positive Prevention Curriculum
  Interventions: Behavioral: Positive Prevention PLUS
- Control (No Intervention): Did not receive any sex-related instruction

INTERVENTIONS:
Behavioral: Positive Prevention PLUS — PP+ has elven 45 minute lessons: (1) Getting Started, (2) Life Planning, (3) Healthy Relationships, (4) Relationship Violence, (5) Family Planning and Contraceptives, (6) Myths and Stereotypes, (7) HIV Disease and AIDS, (8) Recognizing and Reducing Risk, (9) Peer and Media Pressures, (10) Human Immunodeficiency Virus (HIV)/Sexually Transmitted Disease (STD) Testing and Community Resources, and (11) Steps to Success.
  Arms: Treatment

SUMMARY:
This study aims to determine if the Positive Prevention PLUS teen pregnancy prevention program has an impact on abstinence, birth control use, and likelihood of becoming pregnant.

DETAILED DESCRIPTION:
A clustered randomized controlled trial (CRCT) was employed where participating high school sites were randomly assigned either to a treatment group that implemented the Positive Prevention PLUS program or a control group. Students completed a self-administered survey at baseline (prior to program implementation) and a 6 month follow-up survey (post program implementation). Eligible students in the sample included all male and female 9th-grade students from 21 high schools enrolled in mandatory 9th-grade health, science, or physical education classes, to which the district assigns students randomly. Of the 7,042 eligible students, 4,267 received parental consent and were enrolled in the study. Outcome variables include initiation of sexual activity, ever been pregnant, and birth control use.

ELIGIBILITY:
Inclusion Criteria:

* Must have parental consent and be in the eligible school sites.

Exclusion Criteria:

-

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 4267 (Actual)
Dates: Start 2013-08; Primary Completion 2014-05 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Ever had sex (Yes/No) | 6 months
  Ever had sex (Yes/No)
Ever been pregnant (Yes/No) | 6 months
  Ever Been Pregnant (or gotten someone pregnant) (Yes/No)
Sex without using birth control in prior 3 months (Yes/No) | 6 months
  Ever had sex without using birth control in prior 3 months (Yes/No)

CONTACTS AND LOCATIONS:
Locations (1):
- CSUSB, San Bernardino, California, United States